CLINICAL TRIAL: NCT06737484
Title: Effect of Topically Applied Olive Oil on Pruritus in Hemodialysis Patients: Pretest-posttest Model With Control Group
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Collaborators: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Kübra Çırak, Lecturer, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: INONU-SBE-KC-01
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2024-12

CONDITIONS: Hemodialysis Patients; Pruritus
Keywords: Hemodialysis; Nursing; Olive Oil; Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Hemodialysis patient with pruritus who will be treated with olive oil
  Interventions: Other: APPLYING TOPICAL OLIVE OIL
- Control group (No Intervention): Hemodialysis patient with pruritus who will not undergo any intervention

INTERVENTIONS:
Other: APPLYING TOPICAL OLIVE OIL — 1. Preparation phase: Before the application, hand hygiene will be provided, materials will be prepared, and the application will be carried out wearing gloves. The patient bed will be prepared, a stretcher cover and a bed protector will be laid. A screen will be used for patient privacy and only the areas to be applied will be opened in order. Itchy areas will be identified. Before starting the application, olive oil will be tested by applying it to a small area on the inside of the patient's arm in case of any allergic reaction.
  2. Application of olive oil: 3 drops of olive oil will be dropped on the itchy areas (excluding the scalp and private areas) for every 25 cm square area and gently spread over the area for 30-60 seconds. Since there is a 5-7 minute absorption period from the skin, the area will be kept open and then a VAS score will be taken.
  3. After the application: The procedure will be marked on the patient follow-up form.
  Arms: Experimental group

SUMMARY:
Pruritus is one of the common symptoms and complaints in hemodialysis patients. The studies reviewed demonstrated that a number of nonpharmacological interventions are effective in relieving pruritus in hemodialysis patients. Among these interventions, moisturizers were found to be highly effective. This clinical trial study was planned considering that the moisturizing and anti-inflammatory properties of olive oil, which will help relieve skin dryness and inflammation that play a role in the pathogenesis of itching, will be effective in solving the itching problem.

Objective: To evaluate the effect of topically applied olive oil on pruritus in hemodialysis patients.

Research Hypotheses:

H0: Topically applied olive oil has no effect on pruritus in hemodialysis patients.

H1: Topically applied olive oil has an effect on pruritus in hemodialysis patients.

Research Type:

The study was planned to be conducted as an experimental study with a pre-test and post-test control group.

Method: The research will be carried out as an experimental study with pre-test and post-test control groups at the KSÜ Health Practice and Research Hospital Hemodialysis Unit and the Turkish Kidney Foundation KSÜ Dialysis Center between 03/02/2025-01/04/2025, the universe will be hemodialysis patients receiving treatment at the hemodialysis unit of the relevant hospital, the sample will consist of a total of 68 patients, 34 experimental and 34 control groups, as a result of power analysis. Data collection tools: Personal Information Form, 5-D Itch Scale, Visual Analog Scale (VAS), Blood values. In the experimental group, olive oil will be applied to the itchy areas of the patients by the researcher on the days they come for hemodialysis, 3 days a week for 2 weeks. Patients will apply olive oil to themselves at home on the days they do not come to dialysis. Pre-test data will be collected from both groups in the first interview. Subsequently, VAS scores of the experimental group will be taken before and after each application. No application will be made to the control group and VAS scores will be taken on the day they come to dialysis. Post-test data will be collected from patients in the experimental and control groups at the end of 2 weeks using the 5-D Itch Scale.

Originality: The absence of any experimental study in the literature using pure olive oil in the management of itching in hemodialysis patients constitutes the strength and originality of the study.

Expected results: Topical olive oil application is expected to be effective in reducing frequent itching complaints in hemodialysis patients.

DETAILED DESCRIPTION:
Chronic renal failure (CRF); is a condition that progresses with a progressive and irreversible decrease in glomerular filtration rate and nephron damage, disrupting the body's endocrine, metabolic and fluid-electrolyte balance. One of the methods of hemodialysis, peritoneal dialysis and kidney transplantation is required in the treatment of chronic renal failure. The most commonly used of these treatment methods is hemodialysis. Hemodialysis is a treatment method that regulates the fluid and solute balance of the blood taken from the patient through a machine containing a membrane. While the impaired renal functions of the patients are partially corrected with hemodialysis, significant complications also occur in many organs and systems. The most common problem related to the skin of these complications is pruritus. Pruritus is an unpleasant sensory and emotional experience that creates a scratching and rubbing sensation on the skin. Pruritus occurs continuously or intermittently in the form of attacks, widespread throughout the body or localized to a certain area, and occurs most frequently in the head, back, limbs and chest. In the pathogenesis of pruritus; skin dryness, proliferation of mast cells in the skin, release of proinflammatory cytokines such as C-Reactive protein (CRP) and interleukin-6 (IL-6), iron deficiency, dialysis-related allergic reactions, hypersensitivity, hypercalcemia, hyperphosphatemia, increased histamine, drugs, neuropathy, opioid system involvement, secondary hyperparathyroidism, increased serum vitamin A levels, serum bile acids, and uremic toxins play a role. Patients experiencing pruritus experience problems such as fatigue, sleep problems, anxiety, depression, social isolation, and aesthetic concerns, which reduce quality of life and personal care and make adaptation to the disease difficult. Secondary skin changes such as lesions, bleeding, delayed wound healing, mechanical skin damage, and infection may be observed in patients due to pruritus. Since the pathophysiology of pruritus is multifactorial and not fully understood, partially effective treatments are available. Studies have shown that many non-pharmacological interventions are effective in relieving pruritus in hemodialysis patients. Among these interventions, moisturizers have been found to be highly effective.

Olive oil is a product that can be easily absorbed from the skin, prevents fluid loss by accelerating the proliferation of the epidermis, increases the softness of the skin and thus moisturizes the skin and gives it elasticity, and has been widely used in skin care in recent years. A compound called oleocanthal, which forms the basis of the effects of nonsteroidal anti-inflammatory drugs and analgesics, has been identified in olive oil. Olive oil contains; antioxidant effect with vitamin E, increasing intravascular endothelial growth factor (VEGF) levels with phenolic compounds, photoprotection, anti-inflammatory, antimicrobial and antiaging effect, moisturizing effect with squalene, cell repair effect with oleic acid and linoleic acid, which has properties similar to breast milk. Since olive oil is completely compatible with human tissue cells thanks to its lipid composition, it is unlikely to cause an allergic reaction when applied to the skin, does not show any cytotoxic effect, and is an easy-to-obtain and use product.

Symptom management has an important place in nursing services. According to studies, pruritus is one of the most common symptoms and complaints in hemodialysis patients, more than half of the patients experience pruritus. Nurses should develop evidence-based solutions to reduce pruritus symptoms in hemodialysis patients and prevent secondary problems that may occur due to pruritus. This study was planned considering that olive oil's moisturizing and anti-inflammatory properties, which will help relieve skin dryness and inflammation, which play a role in the pathogenesis of pruritus, will be effective in solving the pruritus problem.

METHOD

Purpose of the Study:

The purpose of the study is to evaluate the effect of topically applied olive oil on pruritus in hemodialysis patients.

Research Hypotheses:

H0: Topically applied olive oil has no effect on pruritus in hemodialysis patients.

H1: Topically applied olive oil has an effect on pruritus in hemodialysis patients.

Research Type:

The study was planned to be conducted as an experimental study with a pre-test and post-test control group.

Time and Place of the Study:

Data were planned to be collected between 03/02/2025-01/04/2025 at the Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital Hemodialysis Unit and the Turkish Kidney Foundation Kahramanmaraş Sütçü İmam University Dialysis Center.

Research Universe and Sample:

The study universe will consist of hemodialysis patients receiving treatment in the hemodialysis unit of the relevant hospital. The study sample; As a result of the power analysis, 34 experimental and 34 control groups will consist of a total of 68 patients (The sample size was calculated at a 95% confidence level using the "G. Power-3.1.9.2" program in the study. As a result of the analysis, the standardized effect size was found to be 0.9911 at the α=0.05 level, based on previous studies, and the minimum sample size was calculated as 56, with 28 in the experimental group and 28 in the control group, with a theoretical power of 0.95. It was decided to select 20% more.). Selection Method:

In order for patients who meet the research criteria not to interact with each other, those who come for dialysis on the same 3 days of the week will be included in the same group. The group coming on Monday-Wednesday-Friday and the group coming on Tuesday-Thursday-Saturday will be separated into experimental and control groups by lottery. After the experimental and control groups are determined, a simple random number table will be used for the patients to be included in the groups. Variables of the Study:

Dependent variables: Pruritus levels of the patients Independent variables: Topical olive oil applied to the patients Control variables: Introductory characteristics and blood values of the experimental and control groups, itching scores, pre-test mean score, VAS scores

Study materials:

Natural extra virgin olive oil: A brand with an acidity level (expression of oleic acid in 100 gr olive oil as a percentage) of at most 0.8% and a peroxide value (these are compounds that emerge during the oxidation of the oil, indicating the degree of deterioration of the oil) of at most 20 meqO2/kg will be used. Natural extra virgin olive oil is obtained only by mechanical and physical means, which does not cause any change in the oil content, and its acidity level is low (High acidity causes the loss of components such as the main phenolic compounds and squalene in the oil) (23).

Plasma glass dropper colored glass bottle 100 ml Powder-free vinyl gloves: made of a material called PVC, does not contain allergenic substances, and does not use natural latex in its production.

Cardboard paper Disposable elastic stretcher cover: 80x220 cm Bed protector cover: 60x90 cm Tape measure 150 cm

Data collection tools:

Personal Information Form, 5-D Itch Scale, Visual Analog Scale (VAS), Blood values.

Nursing Intervention Protocol (Olive Oil Application Stages):

Patients will be informed about the properties of olive oil and the benefits of its topical application, will be informed about the study, will have them sign an informed consent form and pre-test data will be collected.

Patients who meet the inclusion criteria and accept the study will be given olive oil; On the days when they come for hemodialysis 3 days a week for 2 weeks, the dialysis process will be started and the researcher will apply it to the pruritus areas (except for the scalp and private areas) within the first 2 hours while the patient stays in bed for the procedure. Patients will apply olive oil to themselves at home on the days they do not come to dialysis.

1. Preparation stage: Hand hygiene will be provided before the application, materials will be prepared, and the application will be made by wearing gloves. The patient bed will be prepared, a stretcher cover and a bed protective cover will be laid. A screen will be used for patient privacy and only the areas where the application will be made will be opened in order. Pruritus areas will be identified.
2. Application of olive oil: 3 drops of olive oil will be applied to the pruritus areas (excluding the scalp and private areas) for every 25 cm square area and spread gently over the area for 30-60 seconds. The area will be kept open since it has an absorption period of 5-7 minutes from the skin and then the VAS score will be taken. The amount applied (3 drops of olive oil for every 25 cm square pruritus area) was determined empirically as the amount required to cover the skin without excessive discharge, since there are no studies conducted according to a specific rule in the literature. In order to determine the 25 cm square area, a piece of cardboard cut as 25 cm square will be used to decide how many drops of olive oil will be applied to the area after the patient shows the pruritus area.
3. After the application: The procedure will be marked on the patient follow-up form. If any changes are seen on the skin, it will be recorded. On the days they do not come to dialysis, patients will be trained to apply 3 drops of olive oil to their itchy areas once a day (at the time it is applied in the clinic) and for 2 weeks for every 25 square cm pruritus area, as done in the clinic. It will be explained that the patient follow-up form created by the researcher should be marked and signed by the patients indicating that it is applied daily. Study materials will be provided to the patients.
4. Patients in the control group will only receive routine nursing care applied in the clinic and no intervention will be applied to these patients by the researcher. It will be stated that itching is monitored and VAS scores will be taken on the days they come for dialysis. At the end of the study, patients in the control group will be informed about the full content of the study, its results and olive oil, and if the research results support the application, olive oil will be applied to patients who want it and olive oil will be given as a gift in a 100 ml plasma glass dropper colored glass bottle for them to use.

Data Collection:

The data of the study will be collected by the researcher by interviewing the patients face to face in the hemodialysis unit of the relevant hospital between 03/02/2025-01/04/2025 for 35-45 minutes, 3 days a week for 2 weeks.

Pre-test data will be collected in the first interview using the Personal Information Form, VAS and 5-D Itching Scale for both groups. Then, VAS scores will be taken before and after each application of the experimental group. No application will be made to the control group and VAS scores will be taken on the days they come to dialysis. Post-test data will be collected using the 5-D Itching Scale for the patients in the experimental and control groups at the end of 2 weeks. The last 6 months of blood values of both groups will be followed up.

Evaluation of data:

Data will be analyzed using SPSS for Windows 25.0 program. Weekly average values of daily measurements will be used in the analysis of VAS scores. In this case, 2 measurement VAS scores and 2 measurement 5-D Itch Scale scores will be available for analysis.

Descriptive statistical methods (number, percentage, min-max values, median, mean, standard deviation) will be used when evaluating the data. Cronbach Alpha values will be calculated to test the reliability of the scales used in the study. Chi-square analysis will be applied to test the homogeneity of the groups in terms of demographic characteristics. Fisher exact test will be applied if the expected frequencies in 2*2 cross tables are less than 5.

The compliance of the scales used in the survey with normal distribution will be determined. The normal distribution of the data used depends on the skewness and kurtosis values being between ±3. Parametric tests will be used in statistical evaluations for scales with normal distribution. In scales with normal distribution, independent t-test will be applied for comparing quantitative data between two groups, and dependent t-test will be applied for comparing two dependent stages.

Non-parametric tests will be used in statistical evaluations for scales without normal distribution. In comparing quantitative data in scales that do not have a normal distribution, the independent Mann Whitney U test will be applied to determine the difference between two groups, and the Wilcoxon test will be applied to compare two dependent stages.

In order to examine the differences between the measurements to be taken every month, the Variance Analysis will be applied to repeated measurements in quantitative variables that comply with the normal distribution. The Friedman test will be applied to examine the differences between repeated measurements for quantitative variables that do not comply with the normal distribution.

Correlation analysis will be applied to test the relationship between numerical variables. In cases where the data have a normal distribution, the Pearson correlation will be applied, and in cases where it does not have a normal distribution, the Spearman correlation will be applied. After the correlation tests, regression analyses will be performed to determine the effect size of the influencing factors.

Statistical significance will be accepted as p<0.05.

Ethical and Legal Aspects of the Research:

Permission was obtained from the "Inonu University Clinical Research Ethics Committee" for the research to be conducted (Date: 05.06.2024, Protocol code of the research: 2024/42). The necessary institutional permission was obtained from the Chief Physician of the Kahramanmaras Sutcu Imam University Health Practice and Research Hospital for the research to be conducted in the Hemodialysis Unit and the Turkish Kidney Foundation Kahramanmaras Sutcu Imam University Dialysis Center. The participants will be informed about the research and the "Informed Consent" principle will be fulfilled, stating that they are free to participate or not in the research, the "Respect for Autonomy" principle, stating that the information of the participants participating in the research will be kept confidential, and written and verbal consent will be obtained. Those who are willing to participate in the research will be included in the scope of the research. Since individual rights must be protected in the research, the Helsinki Declaration of Human Rights will be adhered to during the study. Since the implementation of the study and the collection of data were conducted by a single researcher and the patients knew which group they were in, blinding will not be possible.

Limitations of the Study:

The study included patients receiving dialysis at the Kahramanmaraş Sütçü İmam University Health Practice and Research Hospital Hemodialysis Unit and the Turkish Kidney Foundation Kahramanmaraş Sütçü İmam University Dialysis Center. Therefore, the results obtained from the study can be generalized to this research group.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the study
* Being over 18 years of age
* Not having a psychiatric problem
* Not having a vision, hearing or speech problem
* Knowing Turkish, being open to communication and cooperation
* Receiving hemodialysis treatment for at least 6 months
* Having three pruritus attacks in the last 2 weeks (each attack lasting 5 minutes or longer) or having intermittent pruritus complaints in the last 6 months
* Not having any open wound, cellulitis, infection, deep vein thrombosis, bleeding, paraplegia or pacemaker in the area to be applied
* Not being allergic to olive oil
* Not applying any not using topical medication, moisturizer etc.
* Not using any traditional complementary alternative treatment method on the pruritus area

Exclusion Criteria:

* Not wanting to participate in the study
* Being under the age of 18
* Having a psychiatric problem
* Having a vision, hearing or speech problem
* Not knowing Turkish, not being open to communication and cooperation
* Not receiving hemodialysis treatment for at least 6 months
* Not defining an pruritus complaint
* Having any open wound, cellulitis, infection, deep vein thrombosis, bleeding, paraplegia or pacemaker in the area to be applied
* Being allergic to olive oil
* Not applying any topical medication, moisturizer etc. to the itchy area product use
* Using any traditional complementary alternative treatment method on the pruritus area

Min Age: 18 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2025-01-27 (Actual); Primary Completion 2025-02-16 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
PRURITUS SEVERITY | 14 DAYS
  It will be evaluated with VAS. Visual Analog Scale (VAS): VAS is a scale developed by Huskisson to convert some values that cannot be measured numerically into numerical form. The two extreme definitions of the parameter to be evaluated are written on both ends of a 10 cm line and the patient is asked to indicate where their own situation fits on this line by drawing a line, putting a dot or pointing. The average of the values obtained for the patients is taken in the evaluation. In this study, a form with a 10 cm long line written on one end as "no pruritus" (0) and "very severe pruritus" (10) on the other will be given to determine the severity of pruritus, and the patient will be asked to mark their own condition on this line. The length of the distance from the place where there is no pruritus to the point marked by the patient will be measured with a standard ruler to determine the severity of the patient's pruritus.
Pruritus complaints | 14 DAYS
  It will be evaluated with the 5-D Itch Scale. The 5-D Itch Scale was developed by Elman, Hyman, Gabriel and Mayo in 2010. The scale consists of 5 sub-dimensions and 8 variables, namely duration, severity, course, area of restriction and distribution of pruritus in the body. It is a scale that provides information about the severity, duration, course of pruritus, its effects on sleep, housework/daily tasks, school/work, social life/leisure activities and the areas where it is seen on the body. The scale can be scored between a minimum of 5 (no itching) and a maximum of 25 points (itching at its highest level). While the duration, severity, course and restriction area of pruritus from the scale sub-dimensions are scored between 1 and 5 points; the distribution in the body is scored by examining a total of 16 body parts and scoring 5 points according to the number of body parts affected, as 0-2=1 point, 3-5=2 points, 6-10=3 points, 11-13=4 points and 14-16=5 points.

CONTACTS AND LOCATIONS:
Locations (1):
- Kahramanmaraş Sütçü İmam Üniversitesi Sağlık Araştırma ve Uygulama Hastanesi, Kahramanmaraş, Kahramanmaraş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided